CLINICAL TRIAL: NCT05959798
Title: High Power Short Duration Ablation Compared to Moderate Power Long Duration Ablation for Pulmonary Vein Isolation: Safety and Acute Procedural Outcome
Brief Title: High Power Short Duration Ablation Compared to Moderate Power Long Duration Ablation for Pulmonary Vein Isolation
Status: Completed | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: POWER PULSE
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High power short duration ablation
  Interventions: Procedure: High power short duration ablation
- Moderate power long duration ablation
  Interventions: Procedure: High power short duration ablation

INTERVENTIONS:
Procedure: High power short duration ablation — Pulmonary vein isolation by high power short duration radiofrequency catheter ablation

SUMMARY:
High Power Short Duration Ablation Compared to Moderate Power Long Duration Ablation for Pulmonary Vein Isolation: safety and acute procedural outcome

ELIGIBILITY:
Inclusion Criteria:

* symptomatic, documented, drug-resistent paroxysmal atrial fibrillation
* effective oral anticoagulation

Exclusion Criteria:

* any prior left atrial ablation procedure
* presence of left atrial thrombus
* secondary atrial fibrillation due to electrolyte imbalance or thyroid disease
* any prior oesophageal or gastric surgery

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with documented paroxysmal atrial fibrillation, not previously treated by left atrial catheter ablation
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Number of reconnected pulmonary veins 20 minutes after ablation in comparison of both ablation groups | Acute endpoint

SECONDARY OUTCOMES:
Time to first documented recurrence of atrial fibrillation after a 6-week blanking period. | 12 months after ablation

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Deisenhofer, Prof. Dr., Principal Investigator — Deutsches Herzzentrum München, Abt. für Elektrophysiologie
Locations (1):
- Deutsches Herzzentrum München, München, Germany

IPD SHARING:
Plan to Share IPD: No